CLINICAL TRIAL: NCT03034343
Title: Effectiveness of a Brief Psychological Mindfulness Based Intervention for the Treatment of Depression in Primary Care: Face-to-face Application, Treatment as Usual and Application Through ICTs
Brief Title: Effectiveness of a Brief Psychological Mindfulness Based Intervention for the Treatment of Depression in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Research Unit in Primary Care of Aragon (Spain) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PI16/0202
Record Dates: First submitted 2017-01-11; First posted 2017-01-27 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Depressive Disorder
Keywords: Mindfulness; Internet program; Depression; Cost-effectiveness
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAU+mindfulness applied face to face (Experimental): 4 sessions of 90 minutes/session Mindfulness based intervention applied in groups of 10-12 people in traditional format. Written material and sound recordings will be offered as support elements. The estimated duration of the face to face program is one month.
  Interventions: Behavioral: Mindfulness
- TAU + Mindfulness ICTs intervention (Experimental): 4 sessions of 60 minutes/session Mindfulness based intervention applied by ICTs (Internet-based program). The online intervention will be individual and interactive, which will be supported by multimedia material (videos, sound recordings, etc.) and will have internet support. The estimated duration of the online program is two months.
  Interventions: Behavioral: Mindfulness
- Usual medical treatment (TAU) (No Intervention): In this group the general practitioner will apply the usual treatment (medication) but there will be no psychological treatment.

INTERVENTIONS:
Behavioral: Mindfulness
  Arms: TAU + Mindfulness ICTs intervention; TAU+mindfulness applied face to face

SUMMARY:
The aim of this study is to assess and compare a mindfulness low-intensity (4 weeks) psychological intervention for the treatment of depression in Primary Care between different groups: a mindfulness intervention applied face to face in group format, a control group that will receive treatment as usual (TAU) consisting of medical treatment and the same mindfulness intervention applied by Information and Communication Technologies (ICTs). The principal hypothesis is that face to face intervention will be more effective than TAU

DETAILED DESCRIPTION:
The aim of this study is to assess and compare a mindfulness low-intensity (4 weeks) psychological intervention for the treatment of depression in Primary Care between different groups: 1) a face-to-face mindfulness intervention in group format (10-12 people/group), 2) a control group which will received primary care TAU (usual medical treatment) and 3) the same mindfulness intervention applied by Information and Communication Technologies (ICTs) (Internet-based program). All participants in the two psychological intervention groups will also receive usual medical treatment managed by their general practitioner. Each group will be composed of 40 participants with a total sample of 120. The principal hypothesis is that face to face intervention will be more effective than TAU. Secondary hypothesis, are: 1) The online computerized program will be more effective than TAU; 2) The differences between face-to-face and online format will be analyzed. Finally, a qualitative study will be conducted in order to analyze the feasibility, acceptance, barriers and causes of drop-outs and success, expectations, experiences and attitudes that could be obstacles or facilitators in the interventions, both in patients and in health professionals. This study will allow us to understand the experiences of depressed patients with these interventions and their differences.

ELIGIBILITY:
Inclusion Criteria:

* Be adult
* Willingness to participate in the study and signing informed consent
* Ability to understand and write Spanish.
* DSM-5 diagnose of Major Depression or Dysthymia, mild or moderate depression expressed as score lower than 14 in the Patient Health Questionnaire (PHQ)
* Duration of depressive symptoms 2 months or more
* To have and to handle the computer and internet

Exclusion Criteria:

* Any diagnose of disease that may affect central nervous system (brain pathology, traumatic brain injury, dementia, etc.),
* Other psychiatric diagnoses or acute psychiatric illness (substance dependence or abuse, history of schizophrenia or other psychotic disorders, eating disorders, etc.), except for anxious pathology or personality disorders
* Any medical, infectious or degenerative disease that may affect mood, presence of delusional ideas or hallucinations consistent or not with mood, and suicide risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | Baseline
Beck Depression Inventory-II | Post-treatment 8 weeks from baseline in 8 weeks intervention group
  In the mindfulness-based intervention applied by ICTs
Beck Depression Inventory-II | post-treatment 4 weeks from baseline in 4 weeks intervention group
  In the mindfulness-based intervention applied face-to-face and TAU group
Beck Depression Inventory-II | Six-months follow-up
Beck Depression Inventory-II | Twelve-months follow-up

SECONDARY OUTCOMES:
Sociodemographic data Gender, age, marital status, education, occupation, economical level | Baseline
Health Survey 12 (SF-12) | Baseline
Health Survey 12 (SF-12) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
  In the mindfulness-based intervention applied by ICTs
Health Survey 12 (SF-12) | Post-treatment 4 weeks from baseline in 4 weeks intervention group
  In the mindfulness-based intervention applied face-to-face and TAU group
Health Survey 12 (SF-12) | Six-months follow-up
Health Survey 12 (SF-12) | Twelve-months follow-up
EuroQol (EQ-5D). Health related quality of life | Baseline
EuroQol (EQ-5D). Health related quality of life | Six-months follow-up
EuroQol (EQ-5D). Health related quality of life | Twelve-months follow-up
Positive and negative affect (PANAS) | Baseline
Positive and negative affect (PANAS) | Post-treatment 8 weeks from baseline in 8 weeks intervention group
  In the mindfulness-based intervention applied by ICTs
Positive and negative affect (PANAS) | Post-treatment 4 weeks from baseline in 4 weeks intervention group
  In the mindfulness-based intervention applied face-to-face and TAU group
Positive and negative affect (PANAS) | Six-months follow-up
Positive and negative affect (PANAS) | Twelve-months follow-up
Five Facets and factors of mindfulness (FFMQ) | Baseline
Five Facets and factors of mindfulness (FFMQ) | Six-months follow-up
Five Facets and factors of mindfulness (FFMQ) | Twelve-months follow-up
Pemberton Happiness Index (PHI) | Baseline
Pemberton Happiness Index (PHI) | Six-months follow-up
Pemberton Happiness Index (PHI) | Twelve-months follow-up
Patient Health Questionnaire-9 | Baseline
Patient Health Questionnaire-9 | Post-treatment 8 weeks from baseline in 8 weeks intervention group
  In the mindfulness-based intervention applied by ICTs
Patient Health Questionnaire-9 | Post-treatment 4 weeks from baseline in 4 weeks intervention group
  In the mindfulness-based intervention applied face-to-face and TAU group
Patient Health Questionnaire-9 | Six-months follow-up
Patient Health Questionnaire-9 | twelve-months follow-up

OTHER OUTCOMES:
Client Service Receipt Inventory (CSRI) | Baseline
  This inventory includes the number of times health services have been used.Collect the sick leave, the number of hospital admissions, the number of times that the person attends an emergency service, number of times that is attended by a healthcare professional and finally collects the medication. There is no maximum or minimum score, it simply provides information.
Client Service Receipt Inventory (CSRI) | Six-months follow-up
  This inventory includes the number of times health services have been used.Collect the sick leave, the number of hospital admissions, the number of times that the person attends an emergency service, number of times that is attended by a healthcare professional and finally collects the medication. There is no maximum or minimum score, it simply provides information.
Client Service Receipt Inventory (CSRI) | Twelve-months follow-up
  This inventory includes the number of times health services have been used.Collect the sick leave, the number of hospital admissions, the number of times that the person attends an emergency service, number of times that is attended by a healthcare professional and finally collects the medication. There is no maximum or minimum score, it simply provides information.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Jaume I, Castellon, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersson G, Titov N. Advantages and limitations of Internet-based interventions for common mental disorders. World Psychiatry. 2014 Feb;13(1):4-11. doi: 10.1002/wps.20083. PMID 24497236
- [Background] Backenstrass M, Joest K, Frank A, Hingmann S, Mundt C, Kronmuller KT. Preferences for treatment in primary care: a comparison of nondepressive, subsyndromal and major depressive patients. Gen Hosp Psychiatry. 2006 Mar-Apr;28(2):178-80. doi: 10.1016/j.genhosppsych.2005.10.001. PMID 16516070
- [Background] Cuijpers P, van Straten A, van Schaik A, Andersson G. Psychological treatment of depression in primary care: a meta-analysis. Br J Gen Pract. 2009 Feb;59(559):e51-60. doi: 10.3399/bjgp09X395139. PMID 19192368
- [Background] Kuyken W, Byford S, Taylor RS, Watkins E, Holden E, White K, Barrett B, Byng R, Evans A, Mullan E, Teasdale JD. Mindfulness-based cognitive therapy to prevent relapse in recurrent depression. J Consult Clin Psychol. 2008 Dec;76(6):966-78. doi: 10.1037/a0013786. PMID 19045965
- [Derived] Lopez-Montoyo A, Quero S, Montero-Marin J, Barcelo-Soler A, Beltran M, Campos D, Garcia-Campayo J. Effectiveness of a brief psychological mindfulness-based intervention for the treatment of depression in primary care: study protocol for a randomized controlled clinical trial. BMC Psychiatry. 2019 Oct 16;19(1):301. doi: 10.1186/s12888-019-2298-x. PMID 31619196
- See also: Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es